CLINICAL TRIAL: NCT00099775
Title: A Randomized Double-Masked Trial of Caspofungin Versus Placebo as Prophylaxis of Invasive Candidiasis in High-Risk Adults in the Critical Care Setting
Brief Title: Caspofungin to Prevent Candidiasis in Adults in Hospital Intensive Care Units
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050057; 05-C-0057
Record Dates: First submitted 2004-12-18; First posted 2004-12-20 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-09

CONDITIONS: Candidiasis
Keywords: Mycoses; Candida; Echinocandin; Immunocompromised Host; Invasive Fungal Infection; Fungal Infection
MeSH Terms: conditions — Candidiasis; Mycoses; Torulopsis; Invasive Fungal Infections | interventions — Caspofungin

INTERVENTIONS:
Drug: Caspofungin

SUMMARY:
This study will examine whether the anti-fungal drug caspofungin can prevent Candida infections in adult patients in intensive care units (ICUs). Caspofungin is approved to treat certain fungal infections, including fungal blood stream infections due to Candida. Because ICU patients are at high risk for Candida, it would be beneficial to have a preventive drug, thereby reducing complications due to infection.

Patients 18 years of age or older who are not pregnant may be enrolled in this study on day 3 or 4 of their ICU admission if they have an expected stay of at least 2 additional days in the ICU.

Participants are randomly assigned to treatment with either caspofungin or placebo (an inactive substance). Before treatment, patients have a medical history and physical examination. Blood and urine tests are done for routine tests and to look for fungal infection. Additional samples that may be collected to test for fungal infection include a rectal swab or stool sample; a wound culture if the patient has a wound, or a sputum culture in patients who have a tube in their throat to help with breathing or are producing sputum.

Patients take caspofungin or placebo once a day for no more than 28 days. In addition, they undergo the following procedures:

* Review of treatment side effects and medicines taken, daily during treatment, 1 week after treatment, and 2 weeks after treatment
* Physical examination once a week, on the last day of treatment, and 1 week after treatment
* Urine test once a week, on the last day of treatment, and 1 week after treatment to look for possible fungal infection
* Blood tests twice a week, on the last day of treatment, 1 week after treatment, and 2 weeks after treatment for laboratory safety tests and to look for fungal infection
* Collection of additional samples (rectal swab or stool sample, wound culture, or sputum sample) once a week, on the last day of treatment, and 1 week after treatment to look for possible fungal infection

DETAILED DESCRIPTION:
This study is designed as a prospective, multi-center randomized double-masked placebo-controlled trial of caspofungin versus placebo for prevention of invasive candidiasis in high-risk adults in the critical care setting. The objective of this study is to evaluate the efficacy of caspofungin as prophylaxis for invasive candidiasis in high-risk ICU subjects by comparing the risk of invasive candidiasis in subjects receiving caspofungin with the risk in those receiving placebo. The secondary objectives are to evaluate the rate of invasive candidiasis in subjects meeting the clinical prediction rule; to prospectively assess the effect of colonization as a risk factor for the development of invasive candidiasis; to evaluate the safety of caspofungin as prophylaxis for invasive candidiasis by summarizing the proportion of subjects who discontinue study therapy because of a drug-related adverse event and the proportion of subjects with one or more drug-related adverse event(s); and to evaluate all-cause mortality. The planned sample size will be 1200 subjects, 1/3 in the control arm and 2/3 in the active treatment arm based on a power of at least 0.8 needed to detect a 50% reduction in incidence from base rate of 11% to 5.5%. High-risk icu subjects greater than or equal to 18 years of age meeting all eligibility criteria with at least 5 days of anticipated ICU stay will be randomized to receive either caspofungin 50 mg/day (70 mg/day for subjects on rifampin) or placebo (normal saline) daily. Caspofungin or placebo will be given intravenously as a single daily dose infused over approximately one hour. Subjects will receive study drug or placebo for the duration on their icu stay, up to a maximum of 28 days.

ELIGIBILITY:
INCLUSION CRITERIA

Subjects who meet all of the following criteria are eligible for enrollment into the study:

Participant, or their legal representative, has signed the informed consent. Sites will follow their institutional review board (IRB) specific guidelines for obtaining informed consent.

Admission to an ICU within the previous 3 days. The subject may be enrolled into this study on Days 3, 4 or 5 of the ICU admission, and MUST HAVE an expected stay of at least 2 additional days in the ICU.

NOTE: The day the subject is admitted to the ICU is Day 1 of ICU Admission. All days are counted in calendar days.

Non-pregnant subjects greater than or equal to 18 years of age. Subjects of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to study entry.

Subject must have at least 1 of the following:

Received at least one dose of any systemic antibiotic on any one of the ICU days before study entry and continue to receive antibiotics at the time of enrollment.

Presence of a central venous catheter at time of enrollment and for 1 additional day during current ICU stay.

And at least 2 of the following:

* Use of total parenteral nutrition on any of Days 1-4 of the ICU admission.
* Any type dialysis on any of Days 1-4 of the ICU admission.
* Any in-patient surgery, done under general anesthesia or epidural block, within the 7 days prior to or on ICU admission. (Excludes placement of vascular catheters.)
* Pancreatitis (documented by CT scan or lipase greater than 1,000 u/L) within the 7 days prior to or on ICU admission.
* More than 1 dose of systemic steroids (prednisone equivalent dose greater than or equal to 20 mg per day) between 7 days prior to and through Day 3 of ICU admission.
* Use of more than 1 dose of other systemic immunosuppressive agents (such as azathioprine, tacrolimus, sirolimus, mycophenolate, monoclonal antibodies, and TNF immunomodulators) within the 7 days prior to or on ICU admission.

EXCLUSION CRITERIA

Subjects who meet any of the following criteria are ineligible for enrollment in the study:

* Allergy or intolerance to caspofungin or any other echinocandin analog.
* Absolute neutrophil count less than 500/mm(3) at study entry or likely to develop such an absolute neutrophil count during the study therapy period.
* A diagnosis of HIV, aplastic anemia, or chronic granulomatous disease.
* Moderate or severe hepatic insufficiency as indicated by a Child-Pugh Score of 7 or higher or cirrhosis due to any cause (Child-Pugh scores are to be calculated only if hepatic insufficiency is suspected.
* Women who are pregnant or breastfeeding.
* Subjects unlikely to survive more than 2 days.
* Subjects who have received a systemic antifungal agent for treatment or prophylaxis within 7 days prior to study entry.
* Subjects with documented active, proven or probable IFI within 7 days prior to study entry.
* Subjects who have previously participated in this study.
* Subjects who have received another investigational agent within 7 days prior to study entry or who are currently receiving another investigational agent.
* Subjects in the ICU greater than 5 days prior to enrollment into this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200
Dates: Start 2004-12; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Mora-Duarte J, Betts R, Rotstein C, Colombo AL, Thompson-Moya L, Smietana J, Lupinacci R, Sable C, Kartsonis N, Perfect J; Caspofungin Invasive Candidiasis Study Group. Comparison of caspofungin and amphotericin B for invasive candidiasis. N Engl J Med. 2002 Dec 19;347(25):2020-9. doi: 10.1056/NEJMoa021585. PMID 12490683
- [Background] Beck-Sague C, Jarvis WR. Secular trends in the epidemiology of nosocomial fungal infections in the United States, 1980-1990. National Nosocomial Infections Surveillance System. J Infect Dis. 1993 May;167(5):1247-51. doi: 10.1093/infdis/167.5.1247. PMID 8486965
- [Background] Banerjee SN, Emori TG, Culver DH, Gaynes RP, Jarvis WR, Horan T, Edwards JR, Tolson J, Henderson T, Martone WJ. Secular trends in nosocomial primary bloodstream infections in the United States, 1980-1989. National Nosocomial Infections Surveillance System. Am J Med. 1991 Sep 16;91(3B):86S-89S. doi: 10.1016/0002-9343(91)90349-3. PMID 1928197